CLINICAL TRIAL: NCT04895059
Title: Study of no Pharmacokinetic Interaction Between Rosuvastatin 20 mg and Ezetimibe 10 mg, Open Design, Randomized, Single Dose, 3x6, Crossove, Healthy Volunteers in Fasting, in Fixed Combination Against Individuals Components Managed
Brief Title: Study of no Pharmacokinetic Interaction Between Rosuvastatin 20mg and Ezetimibe10mg, Fixed Dose vs Individual Components
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RSEZ-25-SIL
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Dyslipidemia; Rosuvastatin; Ezetimibe; Cholesterol
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Rosuvastatin / Ezetimibe fixed dose (Experimental): In fixed dose Pharmaceutical Form: Tablets Dosage: 20 mg / 10 mg Administration way: oral
  Interventions: Drug: Rosuvastatin (20mg) /Ezetimibe (10mg) in fixed dose
- Group B: Rosuvastatin (Crestor®) (Active Comparator): Pharmaceutical Form: Tablets Dosage: 20 mg Adminstration wat: Oral
  Interventions: Drug: Rosuvastatin 20mg
- Group C: Ezetimibe (Ezetrol®) (Active Comparator): Pharmaceutical Form: Tablets Dosage: 10 mg Adminstration wat: Oral
  Interventions: Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Rosuvastatin (20mg) /Ezetimibe (10mg) in fixed dose — Form: Tablets Dosage: 20 mg Adminstration way: Oral
  Other Names: ROSU/EZET
  Arms: Group A: Rosuvastatin / Ezetimibe fixed dose
Drug: Rosuvastatin 20mg — Pharmaceutical Form: Tablets Dosage: 20 mg Adminstration way: Oral
  Other Names: ROSU (Crestor®)
  Arms: Group B: Rosuvastatin (Crestor®)
Drug: Ezetimibe 10mg — Pharmaceutical Form: Tablets Dosage: 10 mg Adminstration way: Oral
  Other Names: EZET (Ezetrol®)
  Arms: Group C: Ezetimibe (Ezetrol®)

SUMMARY:
Monocentric study of no pharmacokinetic interaction between rosuvastatin 20 mg and ezetimibe 10 mg. An open design, randomized, single dose with three periods, six sequences and crossed, in healthy volunteers with fasting conditions, managed in fixed dose combination (Sponsor Laboratorios Silanes S.A. de C.V.) versus individual components managed by separated (Crestor®, product of Astrazeneca, S.A. de C.V and Ezetrol®. product of Undra S.A. de C.V.)

DETAILED DESCRIPTION:
To statistically compare the bioavailability of rosuvastatin 20 mg and ezetimibe 10 mg in a pharmacokinetic non-interference study, after single-dose oral administration of a product with the fixed combination of active ingredients with respect to the individual components administered separately in healthy volunteers fasting. In the same way, the safety of the presentations will be evaluated based on the registry of adverse events at the end of the three study periods. The classic 90% confidence intervals will be determined for the intra-individual ratios (test / reference) of the main parameters AUC0-t, AUC0-inf, Cmax for rosuvastatin and ezetimibe.

ELIGIBILITY:
Inclusion Criteria:

* The body mass index of the subjects should be between 18.0-27.0 according to Quetelet.
* Women of childbearing age should have a family planning method (including barrier methods, non-hormonal intrauterine devices or bilateral tubal obstruction) or practice abstinence as a lifestyle during the development of the clinical study.
* Volunteers must be healthy, a criterion determined by the results of a complete medical history carried out by the doctors of the Clinical Research site and the laboratory and cabinet studies carried out in certified Clinical Laboratories.
* The limits of variation allowed within normality in the selection visit will be: blood pressure (sitting) from 90 to 130 mmHg systolic and 60 to 90 mmHg diastolic, heart rate between 50 and 100 beats per minute and respiratory rate between 14 and 20 breaths per minute according to current SOP with code CLI-DES-008 " Measure vital sign".
* The vital signs will be taken after 5 minutes of rest in the sedent position.
* The laboratory and office tests that were carried out for the inclusion of the subjects to the study will be: 1. Complete hematic biometry with differential count: Leukocytes, erythrocytes, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean concentration of corpuscular hemoglobin, distribution width of erythrocytes, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils. 2.27-element blood chemistry: glucose, urea, BUN, creatinine, BUN / creatinine ratio, uric acid, cholesterol, HDL cholesterol, triglycerides, LDL cholesterol, non-HDL cholesterol, atherogenic index, total proteins, albumin, globulins, A / ratio G, total bilirubin, direct bilirubin, indirect bilirubin, TGO, TGP, total alkaline phostatase, gamma-glutamyltranspeptidase, DHL, iron, calcium sodium, potassium and chlorine. 3.General urine test. Physical examination (color, appearance, density); chemical test (pH, leukocytes, nitrites, proteins, glucose, ketones, bilirubin, urobilinogen, hemoglobin); microscopic examination (leukocytes, erythrocytes, dysformic erythrocytes, casts, crystals, pavement cells, renal tubular cells, mucoid networks, bacteria and yeasts. 4. Hepatitis B and C test: HBV surface antigen and anti-HCV antibody. 5. HIV test: Anti-HIV 1 and 2 antibodies. 6. VDRL test. 7. Urine drug abuse test at screening visit and approximately 12 hours prior to drug administration. 8. Online alcohol detection test approximately 12 hours prior to drug admission. 9. Serum pregnancy test at screening visit and urine pregnancy test (qualitative) approximately 12 hours before drug administration. 10. 12-lead electrocardiogram (valid for no more than 3 months).

Exclusion Criteria:

* Volunteers with a history of cardiovascular, neurological (uncontrolled seizures), kidney (severe kidney failure), liver (liver failure, active liver disease or increased transaminases that exceed three times the upper limit of normal), pulmonary, muscular (myopathies) ), rhabdomyolysis, hereditary muscle disorders), metabolic, gastrointestinal including constipation, neurological, endpocrine (diabetes mellitus, hypothyroidism), hematopoietic or any type of anemia, mental illness or other organic abnormalities. As well as those who have had a muscle trauma within the 21 days prior to the study.
* Volunteers who require any medication during the course of the study other than the medication being studied.
* Volunteers with a history of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer.
* History of hereditary galactose intolerance, Lapp lactase deficiency, or glucose or galactose malabsorption.
* Volunteers who have been exposed to medications known as liver enzyme inducers or inhibitors or who have taken potentially toxic medications within 30 days prior to the start of the study.
* Volunteers who have received any medications, including vitamins (with or without a prescription) or herbal remedies 30 days (or 7 half-lives) prior to the start of the study.
* Current or recent use of fibrates, niacin, cyclosporine, and protease inhibitors.
* History of muscle toxicity with another HMG-CoA inhibitor or fibrates.
* Volunteers who have been hospitalized for any problem during the six months prior to the start of the study.
* Subjects allergic to any medicine, food or substance. Subjects who have ingested alcohol and / or carbonated and / or xanthine-containing beverages (coffee, tea, cocoa, chocolate, mate, cola soft drinks) or who have ingested charcoal-grilled food or grapefruit juice within 10 hours prior to the start of the hospitalization period, or subjects who smoked tobacco within 10 hours prior to the start of the study.
* Subjects who have donated or lost 450 ml or more of blood within the 60 days prior to the start of the study.
* Subjects with a history of abuse and dependence on alcohol or psychoactive substances.
* Volunteers requiring a special diet for any reason, for example vegetarian.
* Incapacity of any kind that makes it impossible for the volunteer to understand the nature, objective and possible consequences of the study.
* Evidence of uncooperative attitude during the study.
* Volunteers with positive drug abuse, pregnancy and / or alcohol testing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration following the treatment (Cmax | Baseline, 0.25, 0.50, 0.75, 1.00. 2.00, 3.00, 4.00, 5.00, 6.00. 7.00, 8.00, 10.00, 14.00, 24.00. 36.00, 48.00. 72.00 and 96.00 hours
  Evaluate the fixed dose pharmacokinetics profile of rosuvastatin/ezetimibe, employing the maximum observed concentration following the treatment (Cmax)
The area under the curve from time zero to the last measurable concentration (AUC 0-t)using the linear trapezoidal linear-interpolation method | Baseline, 0.25, 0.50, 0.75, 1.00. 2.00, 3.00, 4.00, 5.00, 6.00. 7.00, 8.00, 10.00, 14.00, 24.00. 36.00, 48.00. 72.00 and 96.00 hours
  Evaluate the fixed dose pharmacokinetics profile of rosuvastatin/ezetimibe, employing the area under the curve from time zero to the last measurable concentration (AUC 0-t)using the linear trapezoidal linear-interpolation method.
The area under the curve from time zero to infinity calculated (AUC 0-inf), | Baseline, 0.25, 0.50, 0.75, 1.00. 2.00, 3.00, 4.00, 5.00, 6.00. 7.00, 8.00, 10.00, 14.00, 24.00. 36.00, 48.00. 72.00 and 96.00 hours
  Evaluate the fixed dose pharmacokinetics profile of rosuvastatin/ezetimibe, employing the area under the curve from time zero to infinity calculated (AUC 0-inf).
Time of the maximum measured concentration (Tmax). | Baseline, 0.25, 0.50, 0.75, 1.00. 2.00, 3.00, 4.00, 5.00, 6.00. 7.00, 8.00, 10.00, 14.00, 24.00. 36.00, 48.00. 72.00 and 96.00 hours
  Evaluate the fixed dose pharmacokinetics profile of Rosuvastatin/ezetimibe, employing time of the maximum measured concentration (Tmax).

SECONDARY OUTCOMES:
Sitting blood pressure (mmHg). | Prior to dosing, at 02.00, 06.00,14.00, 24.00, 36.00, 48.00, 72.00 and 96.00 hours
  The sitting blood pressure was measured and registered at case format report throughout the study.
Pulse rate (p/m). | Prior to dosing, at 02.00, 06.00,14.00, 24.00, 36.00, 48.00, 72.00 and 96.00 hours
  The pulse rate was measured and registered at case format report throughout the study.
Respiratory rate (rr). | Prior to dosing, at 02.00, 06.00,14.00, 24.00, 36.00, 48.00, 72.00 and 96.00 hours
  The respiratory rate was measured and registered at case format report throughout the study.
Axillary-body temperature (°C). | Prior to dosing, at 02.00, 06.00,14.00, 24.00, 36.00, 48.00, 72.00 and 96.00 hours
  The axillary-body temperature was measured and registered at case format report throughout the study.
Adverse events | 96 hours
  Any adverse event were classified by severity, treatment and its relationship with the study drug was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Araceli G Medina Nolasco, M.D, Principal Investigator — Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V.
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chu NN, Chen WL, Xu HR, Li XN. Pharmacokinetics and safety of ezetimibe/simvastatin combination tablet: an open-label, single-dose study in healthy Chinese subjects. Clin Drug Investig. 2012 Dec;32(12):791-8. doi: 10.1007/s40261-012-0013-5. PMID 23109219
- [Background] Fellstrom BC, Jardine AG, Schmieder RE, Holdaas H, Bannister K, Beutler J, Chae DW, Chevaile A, Cobbe SM, Gronhagen-Riska C, De Lima JJ, Lins R, Mayer G, McMahon AW, Parving HH, Remuzzi G, Samuelsson O, Sonkodi S, Sci D, Suleymanlar G, Tsakiris D, Tesar V, Todorov V, Wiecek A, Wuthrich RP, Gottlow M, Johnsson E, Zannad F; AURORA Study Group. Rosuvastatin and cardiovascular events in patients undergoing hemodialysis. N Engl J Med. 2009 Apr 2;360(14):1395-407. doi: 10.1056/NEJMoa0810177. Epub 2009 Mar 30. PMID 19332456
- [Background] Glynn RJ, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Ridker PM. A randomized trial of rosuvastatin in the prevention of venous thromboembolism. N Engl J Med. 2009 Apr 30;360(18):1851-61. doi: 10.1056/NEJMoa0900241. Epub 2009 Mar 29. PMID 19329822
- [Background] Kanazawa I, Yamaguchi T, Yamauchi M, Sugimoto T. Rosuvastatin increased serum osteocalcin levels independent of its serum cholesterol-lowering effect in patients with type 2 diabetes and hypercholesterolemia. Intern Med. 2009;48(21):1869-73. doi: 10.2169/internalmedicine.48.2645. Epub 2009 Nov 2. PMID 19881236
- [Background] Kim KJ, Kim SH, Yoon YW, Rha SW, Hong SJ, Kwak CH, Kim W, Nam CW, Rhee MY, Park TH, Hong TJ, Park S, Ahn Y, Lee N, Jeon HK, Jeon DW, Han KR, Moon KW, Chae IH, Kim HS. Effect of fixed-dose combinations of ezetimibe plus rosuvastatin in patients with primary hypercholesterolemia: MRS-ROZE (Multicenter Randomized Study of ROsuvastatin and eZEtimibe). Cardiovasc Ther. 2016 Oct;34(5):371-82. doi: 10.1111/1755-5922.12213. PMID 27506635
- [Background] Lorgelly PK, Briggs AH, Wedel H, Dunselman P, Hjalmarson A, Kjekshus J, Waagstein F, Wikstrand J, Janosi A, van Veldhuisen DJ, Barrios V, Fonseca C, McMurray JJ; CORONA Study Group. An economic evaluation of rosuvastatin treatment in systolic heart failure: evidence from the CORONA trial. Eur J Heart Fail. 2010 Jan;12(1):66-74. doi: 10.1093/eurjhf/hfp172. PMID 20023047
- [Background] McKenney JM. Efficacy and safety of rosuvastatin in treatment of dyslipidemia. Am J Health Syst Pharm. 2005 May 15;62(10):1033-47. doi: 10.1093/ajhp/62.10.1033. PMID 15901588
- [Background] Nakano T, Inoue I, Takenaka Y, Ono H, Katayama S, Awata T, Murakoshi T. Ezetimibe Promotes Brush Border Membrane-to-Lumen Cholesterol Efflux in the Small Intestine. PLoS One. 2016 Mar 29;11(3):e0152207. doi: 10.1371/journal.pone.0152207. eCollection 2016. PMID 27023132
- [Background] Leiter LA, Betteridge DJ, Farnier M, Guyton JR, Lin J, Shah A, Johnson-Levonas AO, Brudi P. Lipid-altering efficacy and safety profile of combination therapy with ezetimibe/statin vs. statin monotherapy in patients with and without diabetes: an analysis of pooled data from 27 clinical trials. Diabetes Obes Metab. 2011 Jul;13(7):615-28. doi: 10.1111/j.1463-1326.2011.01383.x. PMID 21332628
- [Background] Takayama T, Hiro T, Yamagishi M, Daida H, Hirayama A, Saito S, Yamaguchi T, Matsuzaki M; COSMOS Investigators. Effect of rosuvastatin on coronary atheroma in stable coronary artery disease: multicenter coronary atherosclerosis study measuring effects of rosuvastatin using intravascular ultrasound in Japanese subjects (COSMOS). Circ J. 2009 Nov;73(11):2110-7. doi: 10.1253/circj.cj-09-0358. Epub 2009 Oct 5. PMID 19801853
- [Background] Yu CC, Lai WT, Shih KC, Lin TH, Lu CH, Lai HJ, Hanson ME, Hwang JJ. Efficacy, safety and tolerability of ongoing statin plus ezetimibe versus doubling the ongoing statin dose in hypercholesterolemic Taiwanese patients: an open-label, randomized clinical trial. BMC Res Notes. 2012 May 23;5:251. doi: 10.1186/1756-0500-5-251. PMID 22621316
- See also: Drungbank. Ezetimibe — http://www.drugbank.ca/drugs/DB00973
- See also: NORMA oficial Mexicana NOM-177-SSA1-2013, Que establece las pruebas y procedimientos para para demostrar que un medicamento es intercambiable. Requisitos a que deben sujetarse los Terceros Autorizados que realicen las pruebas de intercambiabilidad — https://www.dof.gob.mx/nota_detalle.php?codigo=5314833&fecha=20/09/2013
- See also: NORMA Oficial Mexicana NOM-220-SSA1-2016, Instalación y operación de la farmacovigilancia. — http://dof.gob.mx/nota_detalle.php?codigo=5490830&fecha=19/07/2017